CLINICAL TRIAL: NCT07224607
Title: A Longitudinal Study Investigating the Effects of Photobiomodulation (PBM) on Cognitive Function and Alzheimer's Disease (AD)-Related Biomarkers in Individuals With Mild Cognitive Impairment (MCI) or Dementia Due to AD
Brief Title: Transcranial Photobiomodulation (tPBM) in Alzheimer's Disease Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Golnaz Yadollahikhales, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00004349
Record Dates: First submitted 2025-11-01; First posted 2025-11-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer's Disease
Keywords: photobiomodulation; PBM; Alzheimer's Disease; Dementia; Mild cognitive impairment; MCI; 1064nm
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active photobiomodulation (Experimental): 1064nm photobiomodulation to be applied for 8 minutes total each session
  Interventions: Device: Photobiomodulation
- Sham (Sham Comparator): only 5 seconds of photobiomodulation, to account for small amount of participants who reported an initial warm sensation upon stimulation
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — 1064nm transcranial photobiomodulation

SUMMARY:
The purpose of this study is to see if a special light treatment, called photobiomodulation, can help people with memory problems such as Mild Cognitive Impairment or Mild Dementia due to Alzheimer's disease. The light is given to the forehead using an FDA-cleared medical device. This device is cleared to provide topical heating to elevate tissue temperature for temporary relief of muscle and joint pain, muscle spasm and stiffness associated with arthritis. It also increases blood circulation and relaxes muscle tissue. This device is being used "off-label," meaning it will be used in a way that is different than its cleared use.

We want to learn whether this light treatment can improve executive function, and whether it changes certain inflammatory and neurodegeneration related signals in the blood. To do this, we will apply the photobiomodulation device to your forehead. We will also ask you questions and give you cognitive tests before and after light treatment. We will also collect blood samples before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form (either by subject or LAR)
* Willingness and ability to comply with all study procedures
* Age 55 to 89 years, inclusive
* Clinical diagnosis of Mild Cognitive Impairment or mild dementia (CDR Global = 0-1; MoCA 16-25) due to probable Alzheimer's disease diagnosis
* Ability to attend in-person sessions at Cedars-Sinai and adhere to weekly visits
* Stable dose of Alzheimer's disease medications (e.g., donepezil, rivastigmine, memantine, galantamine) for at least 4 weeks prior to enrollment, if applicable

Exclusion Criteria:

* Presence of significant neurological conditions other than AD (e.g., epilepsy, Parkinson, etc.)
* History of Seizures
* If patient holds neuroimaging showing space-occupying lesions
* If patient holds imaging with Fazekas greater than or equal to 3, more than 2 lacunar infarcts, and/or more than 5 microhemorrhages
* Current pregnancy or lactation (although unlikely in this population)
* Participation in another clinical trial or investigational drug within the past 30 days
* Active use of illicit substances or non-prescribed psychoactive drugs within the past 30 days.
* Severe dementia due to Alzheimer's disease or another etiology
* Physical or mental impairment that prevents the participant from complying with the cognitive testing battery.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
NIH Toolbox | Baseline measurements will be performed prior to intervention, post-treatment (week 5), and lastly at the 3-month follow-up visit
  Three validated NIH Toolbox tasks:
  1. Dimensional Change Card Sort Task (measure of cognitive flexibility)
  2. Flanker Inhibitory Control and Attention Test (a measure of inhibitory control and selective attention),
  3. Visual Reasoning Test (non-verbal and visual reasoning)

SECONDARY OUTCOMES:
Glial Fibrillary Acidic Protein (GFAP) | Will be performed at baseline and at 3 month follow up
  Plasma GFAP concentration (pg/ml) measure using the S-PLEX Assay
Neurofilament Light Chain (NfL) | Baseline and 3-month follow up
  Plasma Neurofilament Light Chain (NfL) concentration (pg/ml) measure using the S-PLEX Assay
Total Tau | Baseline and 3-month follow up
  Plasma total tau concentration (pg/ml) measure using the S-PLEX Assay
Interferon-γ (IFN-γ) | Baseline and 3-month follow up
  Plasma GFAP concentration (pg/ml) measure using the V-PLEX Assay
Interleukin-1β (IL-1β) | Baseline and 3-month follow up
  Plasma IL-1β concentration measured using the V-PLEX assay
Tumor Necrosis Factor-α (TNF-α) | Baseline and 3-month follow up
  Plasma TNF-α concentration (pg/ml) measured using the V-PLEX assay

CONTACTS AND LOCATIONS:
Overall Officials: Golnaz Yadollahikhales, MD, Principal Investigator — Cedars Siinai Medical Center Department of Neurology
Locations (1):
- CSMC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication all IPD and supporting information will be made available
Access Criteria: All information regarding participants' data on primary and secondary outcome measures that will be used in publication

REFERENCES:
- [Background] Zhu G, Tong Q, Ye X, Li J, Zhou L, Sun P, Liang F, Zhong S, Cheng R, Zhang J. Phototherapy for Cognitive Function in Patients With Dementia: A Systematic Review and Meta-Analysis. Front Aging Neurosci. 2022 Jun 30;14:936489. doi: 10.3389/fnagi.2022.936489. eCollection 2022. PMID 35847661
- [Background] Luo G, Zhang J, Song Z, Wang Y, Wang X, Qu H, Wang F, Liu C, Gao F. Effectiveness of non-pharmacological therapies on cognitive function in patients with dementia-A network meta-analysis of randomized controlled trials. Front Aging Neurosci. 2023 Mar 2;15:1131744. doi: 10.3389/fnagi.2023.1131744. eCollection 2023. PMID 36967820
- [Background] Chan AS, Lee TL, Yeung MK, Hamblin MR. Photobiomodulation improves the frontal cognitive function of older adults. Int J Geriatr Psychiatry. 2019 Feb;34(2):369-377. doi: 10.1002/gps.5039. Epub 2018 Dec 10. PMID 30474306
- [Background] Su M, Nizamutdinov D, Liu H, Huang JH. Recent Mechanisms of Neurodegeneration and Photobiomodulation in the Context of Alzheimer's Disease. Int J Mol Sci. 2023 May 25;24(11):9272. doi: 10.3390/ijms24119272. PMID 37298224
- [Background] Gonzalez-Lima, F. (2021). Neuroprotection and Neurocognitive Augmentation by Photobiomodulation. In: Opris, I., A. Lebedev, M., F. Casanova, M. (eds) Modern Approaches to Augmentation of Brain Function. Contemporary Clinical Neuroscience. Springer, Cham. https://doi.org/10.1007/978-3-030-54564-2_9
- [Background] Vargas E, Barrett DW, Saucedo CL, Huang LD, Abraham JA, Tanaka H, Haley AP, Gonzalez-Lima F. Beneficial neurocognitive effects of transcranial laser in older adults. Lasers Med Sci. 2017 Jul;32(5):1153-1162. doi: 10.1007/s10103-017-2221-y. Epub 2017 May 2. PMID 28466195
- [Background] Boyer D, Hu A, Warrow D, Xavier S, Gonzalez V, Lad E, Rosen RB, Do D, Schneiderman T, Ho A, Munk MR, Jaffe G, Tedford SE, Croissant CL, Walker M, Ruckert R, Tedford CE. LIGHTSITE III: 13-Month Efficacy and Safety Evaluation of Multiwavelength Photobiomodulation in Nonexudative (Dry) Age-Related Macular Degeneration Using the Lumithera Valeda Light Delivery System. Retina. 2024 Mar 1;44(3):487-497. doi: 10.1097/IAE.0000000000003980. PMID 37972955